CLINICAL TRIAL: NCT04369586
Title: A Single Center, Double-blinded, ,Placebo-controlled Phase I Clinical Trial in Healthy Volunteer to Evaluate Tolerance and Pharmacokinetics of Meplazumab of Injection
Brief Title: A Phase I Clinical Trial of Meplazumab in Healthy Volunteer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MPZ-I-01
Record Dates: First submitted 2020-04-24; First posted 2020-04-30 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — meplazumab; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- meplazumab dose 1 (Experimental): 0.06mg/kg for single dose
  Interventions: Drug: meplazumab for injection; Drug: Placebo
- meplazumab dose 2 (Experimental): 0.12mg/kg for single dose
  Interventions: Drug: meplazumab for injection; Drug: Placebo
- meplazumab dose 3 (Experimental): 0.2mg/kg for single dose
  Interventions: Drug: meplazumab for injection; Drug: Placebo
- meplazumab dose 4 (Experimental): 0.3mg/kg for single dose
  Interventions: Drug: meplazumab for injection; Drug: Placebo
- meplazumab dose 5 (Experimental): 0.42mg/kg for single dose
  Interventions: Drug: meplazumab for injection; Drug: Placebo
- meplazumab dose 6 (Experimental): 0.56mg/kg for single dose
  Interventions: Drug: meplazumab for injection; Drug: Placebo
- meplazumab multiple dose (Experimental): 0.3mg/kg for double doses, 1 dose/week
  Interventions: Drug: meplazumab for injection; Drug: Placebo

INTERVENTIONS:
Drug: meplazumab for injection — single dose: 6 dose level, multiple dose: 0.3mg/kg/dose
Drug: Placebo — placebo

SUMMARY:
This is a single center, double-blinded, placebo-controlled phase I clinical trail in healthy volunteer of meplazumab for injection. The primary objective of this phase I trial is to evaluate the safety, tolerability, pharmacokinetic characteristics and occupancy characteristics of peripheral blood cell receptors of meplazumab in healthy volunteer, and provide a reference for the dosage of meplazumab in phase II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 18≤age≤50 years, males or females;
* body weight ≥50 kg, body mass index (BMI) should be within 19.0 and 24.0 (both ends included),
* Vital signs, physical examination, laboratory examination (blood routine, urine routine, blood biochemical, coagulation, etc.) and electrocardiogram are within the normal range, or beyond the normal range, but the researchers determined that the abnormality has no clinical significance (NCS).
* No bad habits, including tobacco addiction (>5 cigarettes per day) or drink addiction (>15 g of alcohol in a day, and more than two days a week for female, or >25 g in a day, and more than two days a week for male; 15 g of alcohol is equivalent to 450 mL beer, 150 mL wine or 50 mL light liquor), no history of drug abuse (defined as the use of illegal drugs);
* No birth plan during the study and within 6 months of completing the test and are willing to use non-hormonal contraceptive measures;
* Have the ability to communicate normally with medical staff and comply with relevant hospital management regulations;
* Understand the study and be willing to participate in the study, and sign an informed consent form. Incompetent subjects, willing and able to comply with all trial requirements.

Exclusion Criteria:

* History of allergies to drugs, food, protein or specific allergies (asthma, rubella, eczema dermatitis, etc.);
* Vital signs, physical examination, routine laboratory tests (blood routine, urine routine, blood biochemistry, coagulation, etc.), 12-lead ECG and other abnormalities and clinical significance;
* Positive for SARS-CoV-2 specific IgM and IgG antibodies test;
* Fever within 3 days before medication (body temperature ≥38.0 ℃);
* Pregnant or lactating women;
* Have received or are participating in other clinical trials within 3 months before the screening;
* Be diagnosed or suspected to have immunodeficiency or autoimmune diseases; undergo immunosuppressive therapy such as anticancer chemotherapy or radiotherapy before the trial, or have received systemic corticosteroid treatment within the past 6 months;
* With a history of acupuncture syncope reaction;
* Positive for HBV surface antigen, anti-HCV antibody, anti-HIV antibody, and syphilis antibody test;
* Tobacco addiction (>5 cigarettes per day) or drink addiction (>15 g of alcohol in a day, and more than two days a week for female, or >25 g in a day, and more than two days a week for male; 15 g of alcohol is equivalent to 450 mL beer, 150 mL wine or 50 mL light liquor), or can not stop smoking and drinking during the study;
* Participated in blood donation or blood loss ≥400mL within 3 months before screening;
* Patients not suitable to participate in this study by the judgment of the investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Incidence rate of treatment-related adverse events as assessed by CTCAE v5.0 | 0-28 days
  Nature, incidence, and severity of AEs/SAEs, and the relationship to meplazumab treatment.

SECONDARY OUTCOMES:
Pharmacokinetic assessments of meplazumab- AUC0-tn | 0-28 days
  AUC0-tn
Pharmacokinetic assessments of meplazumab- AUC0-∞ | 0-28 days
  AUC0-∞
Pharmacokinetic assessments of meplazumab-half life time | 0-28 days
Pharmacokinetic assessments of meplazumab-Cmax | 0-28 days
  Maximum observed plasma concentration of meplazumab (Cmax)

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of the Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No